CLINICAL TRIAL: NCT05884996
Title: Kabat Training Program in Diagonal Pattern With Elastic Bands for Shoulder in Amateur Swimmers. A Randomized Controlled Clinical Trial
Brief Title: Kabat Training Program With Elastic Bands for Shoulder in Amateur Swimmers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: THERA2020
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Swimming; Proprioceptive Neuromuscular Facilitation; Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF training (Experimental): kabat training with elastic bands for 8 weeks 2 times a week before swimming training. 3 series of 10-15 repetitions will be performed
  Interventions: Other: PNF training
- Control group (No Intervention): swimming training 2 times a week

INTERVENTIONS:
Other: PNF training — Resistance training with elastic bands in diagonals of PNF
  Arms: PNF training

SUMMARY:
It has been shown that 90% of swimmers experience shoulder pain at some point in their career. During the macrocycle, swimmers present significant alterations in the muscular balance between external and internal rotators of the shoulder: the IR assumes much prominence in strength levels and RE goes progressively weaker.

furthermore, all overhead athletes (such as swimmers) present a glenohumeral Internal Rotation Deficit and an increase in External Rotation.

The objective of this study is to propose an exercise with an elastic band aimed to strengthening the RE of the shoulder to analyze the effects on the muscular balance between IR and RE. In addition, the effect caused in the limitation of internal rotation is going to be studied

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Swimmers minimum 2 times per week

Exclusion Criteria:

* Acute infection
* Shoulder pathology
* Neer and Hawkins-Kennedy test positive

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
change in ROM external rotation of the shoulder in degrees | Change from Baseline at 8 weeks
  Range of motion in external rotation of the shoulder in 90º of abduction measured with goniometry in degrees
change in ROM internal rotation of the shoulder in degrees | Change from Baseline at 8 weeks
  Range of motion in internal rotation of the shoulder in 90º of abduction measured with goniometry in degrees
change in external rotation isometric strength of the shoulder in newton | Change from Baseline at 8 weeks
  isometric strength in external rotation of the shoulder measured with pressure dynamometer in newton
change in internal rotation isometric strength of the shoulder in newton | Change from Baseline at 8 weeks
  isometric strength in internal rotation of the shoulder measured with pressure dynamometer in newton
change in scapular displacement in maximum flexion in centimeters | Change from Baseline at 8 weeks
  horizontal distance covered by the inferior angle of the scapula measured with PALM in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: José A Del Blanco, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT05884996/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT05884996/ICF_001.pdf